CLINICAL TRIAL: NCT02234739
Title: Efficacy and Safety of Voriconazole for Treatment of Invasive Pulmonary Aspergillosis Secondary to COPD: a Multi-center Prospective，Open Cohort Study (VIA-COPD)
Brief Title: Voriconazole for IPA in Chinese Patients With COPD
Acronym: VIA-COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Red Cross Hospital, Hangzhou, China (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Zhejiang Provincial People's Hospital (Other); First People's Hospital of Hangzhou (Other); Second People's Hospital of Hangzhou (Unknown); The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); Ningbo People's Hospital (Unknown); Xiaoshan People's Hospital (Other); Xiaoshan Hospital (Unknown); The First People's Hospital of Huzhou (Other)
Responsible Party: Principal Investigator, caichuang, professor, Red Cross Hospital, Hangzhou, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hangzhou Red Cross Hospital
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Invasive Pulmonary Aspergillosis; COPD
Keywords: voriconazole; COPD; invasive pulmonary aspergillosis; efficacy; safety
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Pulmonary Disease, Chronic Obstructive | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active treatment (Experimental): Chinese patients with invasive pulmonary aspergillosis treated by voriconazole, who has COPD as underlying condition
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — 2-week long intravenous instillation of voriconazole
  Other Names: Vfend

SUMMARY:
voriconazole is recommended as first-line therapy for invasive pulmonary aspergillosis, however the efficacy and safety of voriconazole for treating invasive pulmonary aspergillosis secondary to COPD is not clear. This study aims to investigate the effectiveness and tolerability of intravenous voriconazole for treatment of invasive pulmonary aspergillosis in Chinese patients with COPD, by monitoring changes in clinical symptoms, eradication of aspergillus, improvement of chest imaging as well as record of possible adverse reactions following 2-week intravenous instillation of voriconazole.

DETAILED DESCRIPTION:
This is a multiple-center open-label clinical trial to study the efficacy and safety of voriconazole for treating invasive pulmonary aspergillosis secondary to COPD in Chinese patients.The primary endpoint is treatment success rate as defined by improvement of symptoms related to invasive pulmonary asperillosis, secondary endpoints include the mortality, the eradication of sputum asperillus and profile of adverse reactions following intravenous instillation of voriconazole.

ELIGIBILITY:
Inclusion Criteria:

* Cases of invasive pulmonary aspergillosis secondary to COPD

Exclusion Criteria:

* Use of voriconazole or itraconazole or amphotericin B or caspofungin or micafungin within 4 weeks prior to enrollment
* Known allergy to voriconazole
* Severe impairment of live or kidney function
* Septic shock
* Unwilling to sign informed consent

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
success rate of voriconazole antifungal treatment | 2-week
  treatment success if defined as improve of symptoms related to invasive pulmonary aspergillosis, such as fever, wheezing, chest pain, dyspnea, and hemoptysis

SECONDARY OUTCOMES:
adverse reactions following voriconazole treatment | 2-week
  any adverse events including complaints, physical signs, or laboratory abnormalities

OTHER OUTCOMES:
all-cause mortality of invasive pulmonary aspergillosis secondary to COPD | 2 week
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Chuang Cai, doctor, Principal Investigator — Red Cross Hospital, Hangzhou, China
Locations (1):
- Hangzhou Red Cross Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Tutar N, Metan G, Koc AN, Yilmaz I, Bozkurt I, Simsek ZO, Buyukoglan H, Kanbay A, Oymak FS, Gulmez I, Demir R. Invasive pulmonary aspergillosis in patients with chronic obstructive pulmonary disease. Multidiscip Respir Med. 2013 Sep 4;8(1):59. doi: 10.1186/2049-6958-8-59. eCollection 2013. PMID 24135224
- [Background] Patel DA, Gao X, Stephens JM, Forshag MS, Tarallo M. US hospital database analysis of invasive aspergillosis in the chronic obstructive pulmonary disease non-traditional host. J Med Econ. 2011;14(2):227-37. doi: 10.3111/13696998.2011.564246. Epub 2011 Mar 9. PMID 21385144
- [Background] Ader F, Bienvenu AL, Rammaert B, Nseir S. Management of invasive aspergillosis in patients with COPD: rational use of voriconazole. Int J Chron Obstruct Pulmon Dis. 2009;4:279-87. doi: 10.2147/copd.s4229. Epub 2009 Aug 3. PMID 19684861
- [Background] Walsh TJ, Anaissie EJ, Denning DW, Herbrecht R, Kontoyiannis DP, Marr KA, Morrison VA, Segal BH, Steinbach WJ, Stevens DA, van Burik JA, Wingard JR, Patterson TF; Infectious Diseases Society of America. Treatment of aspergillosis: clinical practice guidelines of the Infectious Diseases Society of America. Clin Infect Dis. 2008 Feb 1;46(3):327-60. doi: 10.1086/525258. No abstract available. PMID 18177225